CLINICAL TRIAL: NCT01700244
Title: Evaluation of a New Cardiac Pacemaker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanostim, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCP004
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation With 2 or 3° AV or Bifascicular Bundle Branch (BBB) Block; Normal Sinus Rhythm With 2 or 3° AV or BBB Block; Sinus Bradycardia With Infrequent Pauses or Unexplained Syncope With EP Findings
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pacemaker (Experimental)
  Interventions: Device: Pacemaker implant

INTERVENTIONS:
Device: Pacemaker implant

SUMMARY:
An evaluation of a safety and performance of a new cardiac pacemaker

ELIGIBILITY:
Inclusion Criteria:

* Subject must have one of the following clinical indications:

  1. Chronic atrial fibrillation with 2 or 3° AV or bifascicular bundle branch block (BBB block) ; or
  2. Normal sinus rhythm with 2 or 3° AV or BBB block and a low level of physical activity or short expected lifespan (but at least one year); or
  3. Sinus bradycardia with infrequent pauses or unexplained syncope with EP findings; and
* Subject ≥18 years of age;
* Subject has life expectancy of at least one year;
* Subject is not enrolled in another clinical investigation;
* Subject is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams;
* Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the EC;
* If female, for 3 months post-operative, subject will actively practice a contraception method, or will practice abstinence, or is surgically sterilized, or is postmenopausal.

Exclusion Criteria:

* Pacemaker dependent;
* Known pacemaker syndrome, have retrograde VA conduction or suffer a drop in arterial blood pressure with the onset of ventricular pacing;
* Hypersensitivity to < 1 mg of dexamethasone sodium phosphate;
* Mechanical tricuspid valve prosthesis;
* Pre-existing pulmonary arterial (PA) hypertension or significant physiologically-impairing lung disease;
* Pre-existing pacing or defibrillation leads;
* Current implantation of an implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT);
* Presence of implanted vena cava filter;
* Presence of implanted leadless cardiac pacemaker;
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Complication rate, where a complication is defined as a serious adverse device effect (SADE) | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sperzel, MD, Principal Investigator — Kerckhoff Clinic
Locations (8):
- Czechia (2):
  - Na Homolce Hospital, Prague, Prague
  - IKEM, Prague
- Germany (3):
  - Kerckhoff Clinic, Bad Nauheim
  - University Hospital Leipzig, Leipzig
  - Heart Hospital Munich, Munich
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - St. Antonius Hospital, Nieuwegein
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Reddy VY, Miller MA, Knops RE, Neuzil P, Defaye P, Jung W, Doshi R, Castellani M, Strickberger A, Mead RH, Doppalapudi H, Lakkireddy D, Bennett M, Sperzel J. Retrieval of the Leadless Cardiac Pacemaker: A Multicenter Experience. Circ Arrhythm Electrophysiol. 2016 Dec;9(12):e004626. doi: 10.1161/CIRCEP.116.004626. PMID 27932427
- [Derived] Knops RE, Tjong FV, Neuzil P, Sperzel J, Miller MA, Petru J, Simon J, Sediva L, de Groot JR, Dukkipati SR, Koruth JS, Wilde AA, Kautzner J, Reddy VY. Chronic performance of a leadless cardiac pacemaker: 1-year follow-up of the LEADLESS trial. J Am Coll Cardiol. 2015 Apr 21;65(15):1497-504. doi: 10.1016/j.jacc.2015.02.022. PMID 25881930
- [Derived] Reddy VY, Knops RE, Sperzel J, Miller MA, Petru J, Simon J, Sediva L, de Groot JR, Tjong FV, Jacobson P, Ostrosff A, Dukkipati SR, Koruth JS, Wilde AA, Kautzner J, Neuzil P. Permanent leadless cardiac pacing: results of the LEADLESS trial. Circulation. 2014 Apr 8;129(14):1466-71. doi: 10.1161/CIRCULATIONAHA.113.006987. Epub 2014 Mar 24. PMID 24664277